CLINICAL TRIAL: NCT04274400
Title: Comorbid Insomnia and Sleep Apnea in Patients Referred to Polysomnography
Brief Title: Comorbid Insomnia and Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Pedro Rodrigues Genta, Associate Professor, University of Sao Paulo General Hospital
Other Study IDs: Insomnia-OSA
Record Dates: First submitted 2020-02-10; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea; Insomnia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred for polysomnography: Patients referred for polysomnography will be classified according to the presence of OSA, insomnia or both.

SUMMARY:
Insomnia and OSA coexist in clinical populations, but the prevalence of comorbid insomnia among OSA patients in the community and risk factors remain poorly known. Little is known about the impact of sleep apnea and insomnia on the quality of life and quality of sleep compared to the presence of one of the sleep disorders alone. Our hypothesis is that the co-existence of OSA and insomnia is high in our community. We also hypothesized that the co-existence of OSA and insomnia promotes greater impairment of quality of life and quality of sleep when compared to the presence of OSA or insomnia alone.

Patients referred to polysomnography will be submitted to 6 questionnaires to assess daytime sleepiness (EPWORTH), insomnia severity index (ISI), anxiety and depression assessment (Beck's anxiety and depression inventory), quality of life assessment(WHOQOL- BREF) and sleep quality assessment (Pittsburgh questionnaire) and they will also be submitted to a polysomnography type III.

It will be calculated the frequency of insomnia, OSA and the comorbidity between insomnia and OSA in the sample. It will be analysed correlations between the insomnia severity index, apnea and hypopnea index, Epworth sleepiness scale, quality of life scale (WHOQOL-BREF), anxiety and depression scale (Beck's anxiety and depression inventory) and Pittsburgh sleep quality scale. Insomnia severity index scores, Epworth sleepiness scale, quality of life scale (WHOQOL-BREF), anxiety and depression scale (Beck anxiety and depression inventory) and Pittsburgh sleep quality scale will be compared according to the presence and absence of OSA and the presence and absence of insomnia and the presence of the comorbidity insomnia and OSA.

ELIGIBILITY:
Inclusion Criteria:

-Individuals who will participate in the task force for the diagnosis of sleep apnea promoted by the State Department of Health in an agreement signed with the Heart Institute

Exclusion Criteria:

* individuals under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who will participate in the task force for the diagnosis of sleep apnea promoted by the State Department of Health in an agreement signed with the Heart Institute
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of obstructive sleeep apnea, insomnia and comorbid sleep apnea and insomnia | 6 months
  Frequency of obstructive sleeep apnea, insomnia and comorbid sleep apnea and insomnia

SECONDARY OUTCOMES:
Correlations between scales: EPWORTH, ISI, Beck's anxiety and depression inventory, WHOQOL-BREF and Pittsburgh questionnaire | 6 months
  Correlations between scales: EPWORTH, ISI, Beck's anxiety and depression inventory, WHOQOL-BREF and Pittsburgh questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Laboratory, Heart Institute, Pulmonary Division, Hospital das Clínicas da Universidade de São Paulo, São Paulo, São Paulo, Brazil